CLINICAL TRIAL: NCT05637164
Title: Second Affiliated Hosptial， School of Medicine, ZheJiang University
Brief Title: Determination of the ED50 and ED95 of Prophylactic Norepinephrine Infusion for Preventing Post-induction Hypotension in Elderly Patients Undergoing Major Abdominal Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2022-0950
Record Dates: First submitted 2022-11-28; First posted 2022-12-05 (Actual); Last update posted 2022-12-05 (Actual); Status verified 2022-11

CONDITIONS: Norepinephrine; Post-induction Hypotension
MeSH Terms: interventions — Norepinephrine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Norepinephrine (Experimental)
  Interventions: Drug: norepinephrine bitartrate

INTERVENTIONS:
Drug: norepinephrine bitartrate — The treatment group will receive a continuous infusion of norepinephrine at the beginning of anesthesia induction until 15 minutes after intubation. The dosage of norepinephrine was decided by the up-and-down sequential allocation method with an initial dose of 0.05 µg/kg/min and a 0.005 µg/kg/min gradient.

SUMMARY:
The goal of this clinical trial is to determine the ED50 and ED95 of prophylactic norepinephrine infusion for preventing post-induction hypotension in elderly patients undergoing major abdominal surgery using up-and-down sequential method . The main question it aims to answer is:

What is the effective concentration of prophylactic norepinephrine infusion for preventing post-induction hypotension in elderly patients.

Participants will receive different concentrations of norepinephrine infusion at the beginning of anesthesia induction until 15 minutes after intubation.

ELIGIBILITY:
Inclusion Criteria:

* aged 65 to 80 years
* Undergoing major abdominal surgery
* American Society of Anesthesiologists (ASA) physical status of I/II/III

Exclusion Criteria:

* Patient refusal
* Severe untreated or uncontrolled hypertension despite medications
* Bradycardia (heart rate < 50 beat per minute)
* Cardiac morbidities, heart block greater than the first degree
* Severe hepatic and renal dysfunction
* hyperthyroidism
* vascular diseases
* BMI>30
* Monoamine oxidase inhibitors were used 2 weeks before surgery

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2023-05-30 (Estimated); Study Completion 2023-05-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of hypotension | 15 minutes after intubation
  less than 80% baseline blood pressure less than 80% baseline blood pressure less than 80% baseline blood pressure

SECONDARY OUTCOMES:
incidence of bradycardia | 15 minutes after intubation
  heart rate less than 50 beat per minute
incidence of reactive hypertension | 15 minutes after intubation
  increased mean arterial pressure by > 20% of the baseline reading

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Zhejiang University Medical College, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No